CLINICAL TRIAL: NCT02283528
Title: A Comparison of Stryker Hybrid Arch Bars Versus Erich Arch Bars for Maxillomandibular Fixation of Mandibular Fractures: A Prospective Randomized Study
Brief Title: A Comparison of Stryker Hybrid Arch Bars
Acronym: Hybrid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Gary F Bouloux MD, DDS, MDSc, FRACDS, FRACDS, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076048
Record Dates: First submitted 2014-10-25; First posted 2014-11-05 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Fracture Mandible
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid (Experimental): Placement of Hybrid arch bars for open or closed reduction of mandible fractures
  Interventions: Device: Stryker Hybrid
- Erich (Active Comparator): Placement of Erich archbars for open or closed reduction of mandible fractures
  Interventions: Device: Erich

INTERVENTIONS:
Device: Stryker Hybrid — Place Hybrid arch bars
  Arms: Hybrid
Device: Erich — Control group is Erich arch bars
  Arms: Erich

SUMMARY:
Patients who sustain a fracture of the lower jaw are typically treated by wiring the teeth together or using small titanium plates and screws to fix the fracture. With either technique the upper and lower teeth are held together to ensure that the fracture is held in the correct position during healing (for closed reduction) or while the plate and screws are applied (for open reduction).

The teeth can be held together using Erich arch bars which are a type of braces that are temporarily wired to the existing teeth. These stay in place for 6 weeks until the fracture has healed even though the patient is able to open his mouth immediately after the surgery is complete. The alternative to the traditional Erich arch bars is a relatively new type of arch bar (Stryker Hybrid) that is screwed to the jaw bone rather than wired to the teeth. The purpose of this study is to compare the two types of arch bars in terms of the speed with which they can be applied as well as any difference in fracture healing

ELIGIBILITY:
Inclusion Criteria:

1. Mandible fracture involving subcondyle, ramus, angle, body, parasymphysis and symphysis
2. Age 18 years - 90 years
3. Ability to give informed consent
4. Minimum 6 weeks follow-up
5. Pre and post-operative panoramic xrays

Exclusion Criteria:

1. Comminuted fractures
2. Infected fractures
3. Previously treated fractures
4. Complete edentulism
5. Gun shot wounds
6. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hybrid | Erich
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hybrid | Erich | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 22 | 20 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 17 | 38
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Time to Place Archbars
Description: Time taken to place archbars
Time Frame: During initial admission and surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hybrid | Erich
Number analyzed (Participants) | 26 | 24
minutes | 14.07 (8.4) | 37.29 (15.1)

2. Secondary Outcome: Number of Participants With Fracture Healing at 6 Weeks
Description: Radiographic healing
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid | Erich
Number analyzed (Participants) | 26 | 24
Participants | 18 | 18

3. Secondary Outcome: Number of Participants With Complications Including Loosening of Archbars, Loosening of MMF, or Damage to Adjacent Teeth and Structures
Description: assess operative and post-operative complications to include loosening of archbars, loosening of MMF if stratified to closed reduction and damage to adjacent teeth and structures
Time Frame: up to 6 weeks post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid | Erich
Number analyzed (Participants) | 26 | 24
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks post baseline
Arm/Group | Hybrid | Erich
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-01-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT02283528/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT02283528/SAP_001.pdf